CLINICAL TRIAL: NCT02431884
Title: Tissue and Bodily Fluid Specimens From Women Presenting to the Reproductive Endocrinology Clinic
Brief Title: Tissue Samples and Bodily Fluid Specimens Banking
Status: Completed | Type: Observational
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01629-XP
Record Dates: First submitted 2015-04-23; First posted 2015-05-01 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Endocrine Disorders of Female Reproductive System
MeSH Terms: interventions — Endomet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — A portion of blood/tissue specimens that will be generated during the participants office visit or surgery.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- body fluids/tissues & history: collect body fluids/tissues & med history from subjects with polycystic ovary syndrome(PCOS), congenital uterine malformations, endocrine malfunctions, endometriosis, and infertility;
  Interventions: Procedure: collect body fluids/tissues & med history

INTERVENTIONS:
Procedure: collect body fluids/tissues & med history — collect tissues/fluids & history
  Other Names: disorders of the ovaries, uterus, endocrine, endometrium

SUMMARY:
The purpose of this study is to collect a portion of blood/tissue specimens that will be generated during the participants office visit or surgery. The investigators are asking whether a small portion of the specimen/s could be set aside and banked for future research purposes. Data originating from participants will be gathered and analyzed in research studies that will help understanding various medical conditions such as polycystic ovary syndrome (PCOS), congenital uterine malformations, endocrine malfunctions, endometriosis, and infertility.

DETAILED DESCRIPTION:
PURPOSE: Women present to the Reproductive Endocrinology clinic with different concerns. These may involve conditions such as pelvic pain, endometriosis, Mullerian anomalies, polycystic ovary syndrome, abnormal uterine bleeding, menopausal symptoms, or infertility. Understanding the meaning of different biologic markers in their blood serum or tissues could help advancing the medical knowledge in the different conditions.

RATIONALE: To understand the meaning of different biologic markers in the patients' blood serum or tissue samples.

POPULATION: Patients identified among all women presenting to the reproductive endocrinology clinic.

Patients may undergo endometrial biopsy or surgery to evaluate their condition. In these instances, the investigators will ask the patients whether a small portion of their specimen/s could be collected and banked for future research purposes.

DESIGN: Prospective blood/tissue collection.

PROCEDURES: A small portion of the patient's blood or tissue specimen collected at the time of a medically indicated blood draw or surgical procedure will be collected and banked for future research purposes. Sample collection will be performed on existing specimens, once the specimens have been obtained for medical indications. No additional procedures will be performed on the patients for research purposes only.

OUTCOME MEASURES: Creation of a blood serum/tissue specimens bank for future clinical research studies.

ELIGIBILITY:
Inclusion Criteria:

* females of childbearing potential experiencing reproductive endocrinology related problems.

Exclusion Criteria:

* male or female not of childbearing potential

Min Age: 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: POPULATION: Patients identified among all women presenting to the reproductive endocrinology clinic.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-01; Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Specimen bank for future clinical research studies | The samples collected during the clinical visit will be preserved and maintained as frozen specimens until the research is performed, which may occur from: within 1 year, and up to 24 years after collection.
  Creation of a blood serum/tissue specimens bank for future clinical research studies.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Detti, M.D., Principal Investigator — Associate Professor, UTennessee Health Science Center
Locations (1):
- Regional One Health Ob-Gyn Clinic, Memphis, Tennessee, United States